CLINICAL TRIAL: NCT00908557
Title: Multicenter RCT to Assess the Impact of Improvements in Lexico-syntactic Readability and Good Practice in Writing on the Comprehension of Written Information Given to Patients Participating in Clinical Trials.
Brief Title: Impact of Readability Improvements on the Comprehension of Written Information Given to Clinical Trial Patients: a RCT
Acronym: LISYCOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Research Center of Grenoble (Unknown); Clinical Research Center of Strasbourg (Unknown); Hôpital Necker-Enfants Malades (Other); Clinical Research Center of Lyon (Unknown); Clinical Research Center of Bichat, Paris (Unknown); Clinical Research Center of Saint-Etienne (Unknown); Clinical Research Center - biotherapy center of Saint-Louis, Paris (Unknown); Clinical Research Center of Clermont-Ferrand (Unknown); Clinical Research Center of Reunion island (Unknown); Clinical Research Center - Biotherapy center of Nantes (Unknown); CIC 1417 Cochin-Pasteur (Other); Pharmacology unit of Créteil (Unknown); Clinical Research Center, Toulouse (Other)
Responsible Party: Principal Investigator, AdministrateurCIC, Pr Jean-Luc CRACOWSKI, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DCIC 08 15
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Comprehension
Keywords: Lexicosyntactic readability improvement; phase II/III trials; ethic; Informed consent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receiving an information and consent form that has been modified using the LISYCOM methods.
  Interventions: Other: readability improvement and good practice redaction
- 2 (Active Comparator): Patients receiving a standard information and consent form.
  Interventions: Other: Control

INTERVENTIONS:
Other: readability improvement and good practice redaction — improvement using Flesch readability index and good practice in redaction of informed consent documents.
  Arms: 1
Other: Control — information based on the classic informed consent document
  Arms: 2

SUMMARY:
The principle objective of this randomised controlled trial is to assess whether an improvement in lexico-syntactic readability combined with adherence to French recommendations for good practice in writing the Information and Consent Form (ICF) given to patients participating in clinical trials, increases their understanding of the information compared to conventional written information, in real (not simulated) conditions.

DETAILED DESCRIPTION:
The quality of written information given to people participating in clinical trials is essential as by law all volunteers have to be informed of a certain number of key elements. Those elements that are necessary to understanding and making a decision as to whether to participate in the trial are presented to the volunteer in the information and consent document (ICD).

Many terms used in the ICD are of necessity medical terms and sometimes difficult to understand for the person who may participate in the study.

Several factors are involved when a reader receives a text, and one of the difficulties of intelligibility can be the lexico-syntactic readability.

The lexico-syntactic readability is the only element of intelligibility that can be readily quantified, using the Flesch-Kincaid index. It is also an element that can be very easily modified without changing the sense of the information.

In the QuIP-3 study, which we performed in 2003, it appeared that the lexico-syntactic readability of ICF is very low, lower than that of texts used in university level classics examinations. Furthermore, there is no correlation between the density of information and readability (QuIP-5 study).

It seems to be necessary to assess the understanding of those participating in clinical trials in terms of logical and cognitive intelligibility (representativeness and interpretability of the information and consent forms). Indeed, a text may be unreadable according to the Flesch score, in lexico-syntactic terms, but perfectly understood and interpreted.

As no questionnaire had been validated in French, we validated the " Questionnaire d'Evaluation de la Compréhension de l'Information Ecrite par les Malades or QECIEM " (Questionnaire measuring patient comprehension of written information) (QuIP-4). This questionnaire can be used to measure both objective and subjective general understanding by a patient to be included in a therapeutic study, irrespective of the pathology.

ELIGIBILITY:
Inclusion Criteria:

* Subject considered suitable to participate in one of the clinical trials selected for the LISYCOM study
* Age > 18 years

Exclusion Criteria:

* Illiteracy or inability to read French
* Neurological deficiency making reading impossible (attention disorders, aphasy, etc)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Sub-score in part A (objective comprehension) of the QECIEM questionnaire of comprehension. | 24 hours

SECONDARY OUTCOMES:
Total score in the QECIEM questionnaire of comprehension. | 24 hours
Sub-scores in part B (subjective comprehension) of questionnaire of comprehension. | 24 hours
Adhesion to proposed clinical trial protocols | end of the study or end of Lisycom
Impact of complementary oral information on the QECIEM scores | 24 hours
Subjective evaluation of readability by the investigator | begin of the study or begin of Lisycom
Number of refusals to sign informed consent form for the proposed trial. | end of the study or end of Lisycom
Score of the QECIEMc | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD, Principal Investigator — Clinical Research Center Grenoble France
Locations (1):
- Clinical Research Center, University Hospital Grenoble, Grenoble, France

REFERENCES:
- [Background] Paris A, Cracowski JL, Ravanel N, Cornu C, Gueyffier F, Deygas B, Guillot K, Bosson JL, Hommel M. [Readability of informed consent forms for subjects participating in biomedical research: updating is required]. Presse Med. 2005 Jan 15;34(1):13-8. doi: 10.1016/s0755-4982(05)83877-1. French. PMID 15685092
- [Background] Paris A, Cracowski JL, Maison P, Radauceanu A, Cornu C, Hommel M. Impact of French 'Comites de Protection des Personnes' on the readability of informed consent documents (ICD) in biomedical research: more information, but not better information. Fundam Clin Pharmacol. 2005 Jun;19(3):395-9. doi: 10.1111/j.1472-8206.2005.00327.x. PMID 15910664
- [Background] Okais C, Paris A, Cracowski JL. [Readability and information density in biomedical research]. Therapie. 2007 Jan-Feb;62(1):17-21. doi: 10.2515/therapie:2007008. Epub 2007 Mar 21. French. PMID 17374343
- [Background] Paris A, Cornu C, Auquier P, Maison P, Radauceanu A, Brandt C, Salvat-Melis M, Hommel M, Cracowski JL. French adaptation and preliminary validation of a questionnaire to evaluate understanding of informed consent documents in phase I biomedical research. Fundam Clin Pharmacol. 2006 Feb;20(1):97-104. doi: 10.1111/j.1472-8206.2005.00391.x. PMID 16448400
- [Background] Paris A, Nogueira da Gama Chaves D, Cornu C, Maison P, Salvat-Melis M, Ribuot C, Brandt C, Bosson JL, Hommel M, Cracowski JL. Improvement of the comprehension of written information given to healthy volunteers in biomedical research: a single-blind randomized controlled study. Fundam Clin Pharmacol. 2007 Apr;21(2):207-14. doi: 10.1111/j.1472-8206.2007.00472.x. PMID 17391294